CLINICAL TRIAL: NCT04103749
Title: Global Prospective Case Series Using a Single-Use Duodenoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: E7156
Record Dates: First submitted 2019-09-20; First posted 2019-09-25 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Exalt DScope 02 (Experimental): Subjects will have a clinically indicated per standard of care ERCP or other duodenoscope-based procedure performed using the Exalt single use duodenoscope study device. Subjects are considered enrolled after completing the study specific informed consent form.
  Interventions: Device: Exalt Model D Single-Use Duodenoscope

INTERVENTIONS:
Device: Exalt Model D Single-Use Duodenoscope — Subjects will have a clinically indicated per standard of care ERCP or other duodenoscope-based procedure performed with the Exalt single use duodenoscope study device.

SUMMARY:
Confirm procedural performance of the ExaltTM Model D Single-Use Duodenoscope in Endoscopic Retrograde Cholangio-Pancreatography (ERCP) and other duodenoscope-based procedures

DETAILED DESCRIPTION:
This study is a prospective, multi-center case series of per standard of care ERCP procedures using a nonsignificant risk single-use duodenoscope. Up to 1000 cases will be included at up to 40 clinical sites. Patients who meet all eligibility criteria will be included and will have a clinically indicated ERCP procedure performed using the study device. Enrolled subjects will be followed for 30 days after their procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study
* Scheduled for a clinically indicated ERCP

Exclusion Criteria:

* Potentially vulnerable subjects, including, but not limited to pregnant women
* Subjects for whom endoscopic techniques are contraindicated
* Patients who are currently enrolled in another investigational study that would directly interfere with the current study, without prior written approval from the sponsor
* Investigator discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2023-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Slivka, MD, PhD, Principal Investigator — University of Pittsburgh Medical Center; Marco Bruno, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (22):
- United States (11):
  - University of California Los Angeles Medical Center, Los Angeles, California
  - University of Chicago, Chicago, Illinois
  - Indianapolis University Hospital, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - North Shore University Hospital, Manhasset, New York
  - Cornell Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- Metro North Hospital and Health Services, Brisbane, Australia
- St. Michael's Hospital - Unity Health, Toronto, Canada
- Institut Paoli-Calmettes, Marseille, France
- Evangelisches Krankenhaus Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany
- Prince of Wales Hospital, Hong Kong, Hong Kong
- India (2):
  - Asian Institute of Gastroenterology, Hyderabad, Telangana
  - Apollo Multispeciality Hospitals, Kolkata, West Bengal
- Humanitas University, Milan, Italy
- Erasmus University Medical Center of Rotterdam, Rotterdam, Netherlands
- Singapore General Hospital, Singapore, Singapore
- Dr. George Mukhari Academic Hospital, Ga-Rankuwa, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruno MJ, Beyna T, Carr-Locke D, Chahal P, Costamagna G, Devereaux B, Giovannini M, Goenka MK, Khor C, Lau J, May G, Muthusamy VR, Patel S, Petersen BT, Pleskow DK, Raijman I, Reddy DN, Repici A, Ross AS, Sejpal DV, Sherman S, Siddiqui UD, Ziady C, Peetermans JA, Rousseau MJ, Slivka A; EXALT Single-use Duodenoscope Study Group. Global prospective case series of ERCPs using a single-use duodenoscope. Endoscopy. 2023 Dec;55(12):1103-1114. doi: 10.1055/a-2131-7180. Epub 2023 Jul 18. PMID 37463599

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exalt DScope 02
Started | 551
Completed | 495
Not Completed | 56

BASELINE CHARACTERISTICS:
Arm/Group | Exalt DScope 02
Number analyzed (Participants) | 551
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (15.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex, Male | 281
  Sex, Female | 269
  Sex, other | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 25
  Netherlands | 25
  Singapore | 25
  Hong Kong | 25
  United States | 276
  Italy | 25
  South Africa | 25
  Australia | 25
  France | 25
  Germany | 25
  India | 50
American Society of Anesthesiology physical status [Count of Participants; unit: Participants] — PI graded physical status of subjects on the ASA scale from I - IV. ASA I being a normal healthy patient to ASA VI being a brain dead patient.
  Participants
    I | 66
    II | 198
    III | 250
    IV | 32
    V | 0
    Not assessed | 5
Relevant gastrointestinal medical history [Number; unit: participants]
  Bile duct stones/gallstones(current) | 168
  Documented biliary or pancreatic stricture, unresolved | 124
  Current immunosuppression (any cause) | 71
  Chronic pancreatitis | 68
  Pancreatic tumor | 63
  Abnormal image finding | 60
  Cholangitis (current) | 53
  Cholangiocarcinoma | 46
  Primary sclerosing cholangitis | 24
  Other gastrointestinal cancer | 22
  Pancreatic stones (current) | 22
  Recurrent cholangitis | 21
  Hepatic tumor | 18
  Hepatitis | 11
  Pancreatic pseudocyst | 9
  Known history of Multidrug-resistant organisms (MDRO) colonization | 2
  Known current MDRO colonization | 2
  Current documented bacterial infection, other than cholangitis | 8
  Other | 146

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful ERCP Procedure
Description: The ability to complete the ERCP procedure for the intended indication(s); outcome reported as "success" or "failure".
  Examples include but are not limited to: biliary stent placement, pancreatic stent placement, sphincterotomy, and clearance of bile duct stones.
Time Frame: Procedure success is assessed at the end of the procedure (within 24 hours on study day 1).
Measure: Count of Participants; unit: Participants
Arm/Group | Exalt DScope 02
Number analyzed (Participants) | 551
Participants | 529

2. Secondary Outcome: Endoscopist Rating
Description: Endoscopist ratings of overall satisfaction with the single-use duodenoscope on a scale of 1 (worst) to 10 (best)
Time Frame: Endoscopists will rate their experience with the Exalt single-use duodenoscope immediately following the completion of the study procedure on study day 1.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Exalt DScope 02
Number analyzed (Participants) | 551
Score on a scale | 8.0 [1.0 to 10.0]

3. Secondary Outcome: Number of Participants With a Crossover From Exalt Single-use Duodenoscope to Reusable Duodenoscope
Description: The need to use a reusable duodenoscope for any task which cannot be adequately performed with the Exalt single-use duodenoscope is considered a crossover.
Time Frame: Incidence of crossover is monitored throughout the procedure (within 24 hours on study day 1).
Measure: Count of Participants; unit: Participants
Arm/Group | Exalt DScope 02
Number analyzed (Participants) | 551
Participants | 37

4. Secondary Outcome: Number of Adverse Events (SAEs) Related to the Device and/or the Procedure
Description: Evaluation of serious adverse events (SAEs) related to the device and/or the procedure through 30 days after the ERCP or other duodenoscope based procedures
Time Frame: SAEs are assessed through 30 days after the procedure.
Measure: Number; unit: Events
Arm/Group | Exalt DScope 02
Number analyzed (Participants) | 551
Events | 46

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | Exalt DScope 02
All-Cause Mortality (participants affected / at risk) | 17/551
Serious Adverse Events (participants affected / at risk) | 85/551
Other Adverse Events (participants affected / at risk) | 75/551
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exalt DScope 02 (N=551)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Duodenal perforation (Gastrointestinal disorders) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 19 (19)
Pneumoretroperitoneum (Gastrointestinal disorders) | 1 (1)
Complication associated with device (General disorders) | 1 (1)
Disease progression (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 6 (6)
Cholecystitis (Hepatobiliary disorders) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Bacteraemia (Infections and infestations) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Post procedural pneumonia (Infections and infestations) | 1 (1)
Pseudomonas peritonitis (Infections and infestations) | 1 (1)
Retroperitoneal abscess (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 5 (5)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 5 (5)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exalt DScope 02 (N=551)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 25 (25)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (8)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 2 (3)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Haemobilia (Hepatobiliary disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Klebsiella infection (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 5 (5)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 2 (2)
Blood pressure increased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Device occlusion (Product Issues) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations include the lack of randomization and the absence of a control group. The enrolled subjects may not be typical of patients at all endoscopy centers. Several investigators participated in the development of the single-use duodenoscope and also received research funding from the study sponsor and from manufacturers of reusable duodenoscopes. Lastly, this study did not address the associated costs or impact on reprocessing services or the environment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the right to discuss or publish trial results without prior review by the Sponsor

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT04103749/Prot_SAP_002.pdf